CLINICAL TRIAL: NCT05263388
Title: A Randomised, Controlled, Assessor-blind, Parallel Groups, Multicentre, Multinational Trial Comparing the Ovarian Response of a Starting Dose of 15 μg Follitropin Delta (REKOVELLE) to a Starting Dose of 225 IU Follitropin Alfa (GONAL-F) in Conventional Regimens in Controlled Ovarian Stimulation in Women Undergoing an Assisted Reproductive Technology Programme
Brief Title: A Trial to Compare the Ovarian Response of REKOVELLE and GONAL-F in Conventional Dosing in Women Undergoing Controlled Ovarian Stimulation
Acronym: ADAPT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000401; U1111-1267-1119 (Other: WHO UTN)
Record Dates: First submitted 2021-11-16; First posted 2022-03-02 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin delta; follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REKOVELLE (Follitropin Delta) (Experimental)
  Interventions: Drug: REKOVELLE (Follitropin Delta)
- GONAL-F (Follitropin Alfa) (Active Comparator)
  Interventions: Other: GONAL-F (Follitropin Alfa)

INTERVENTIONS:
Drug: REKOVELLE (Follitropin Delta) — REKOVELLE administered as single daily subcutaneous injections in the abdomen. The starting dose of REKOVELLE was 15 μg fixed for the first four stimulation days. Dose adjustments could be implemented on the day of starting the gonadotropin-releasing hormone (GnRH) antagonist (stimulation day 5 or day 6) or later, could occur no more frequently than every second day. At each dose adjustment, the daily REKOVELLE dose could be increased or decreased by 5 μg based on the participant's response. The minimum REKOVELLE dose was 5 μg and the maximum REKOVELLE was 20 μg. Participants could be treated for a maximum of 20 days.
  Arms: REKOVELLE (Follitropin Delta)
Other: GONAL-F (Follitropin Alfa) — GONAL-F administered as single daily subcutaneous injections in the abdomen. The starting dose of GONAL-F was 225 IU fixed for the first four stimulation days. Dose adjustments could be implemented on the day of starting the GnRH antagonist (stimulation day 5 or day 6) or later, could occur no more frequently than every second day. At each dose adjustment, the daily GONAL-F dose could be adjusted by 75 IU based on the participant's response. The minimum GONAL-F dose was 75 IU and the maximum GONAL-F dose was 300 IU. Participants could be treated for a maximum of 20 days.
  Arms: GONAL-F (Follitropin Alfa)

SUMMARY:
Hormone preparations like REKOVELLE and GONAL-F are used to make the body produce multiple egg sacs, allowing more eggs to be collected from women undergoing infertility treatment.

The main purpose of this trial is to see how many eggs are produced with a starting dose of 15 µg REKOVELLE compared to a starting dose of 225 IU GONAL-F. This research is intended to provide more knowledge about REKOVELLE, including the doses given in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women aged 18-40 years
* Diagnosed with tubal infertility, unexplained infertility, mild endometriosis (stage I/II) or partners with decreased sperm quality
* Medically eligible for in vitro fertilization (IVF) and/or intracytoplasmic sperm injection (ICSI)
* Infertility for at least one year for participants ≤ 37 years or for at least 6 months for participants ≥ 38 years
* Regular menstrual cycles of 21-35 days.

Exclusion Criteria:

* Known condition of not functioning ovaries
* Known advanced endometriosis (stage III/IV)
* Considered unsuitable for controlled ovarian stimulation with a dosing regimen corresponding to approximately 225 IU/day gonadotropin, as judged by the investigator
* History of previous episode of OHSS or exuberant ovarian response to gonadotropins, and polycystic ovarian syndrome
* Any known hormonal or metabolic abnormalities which can compromise participation in the trial
* Known tumors of the ovary, breast, uterus, adrenal gland, pituitary or hypothalamus

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 302 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (16):
- Austria (2):
  - Ferring Investigational Site, Wals-Seizenheim, Salzburg
  - Ferring Investigational Site, Vienna
- France (2):
  - Ferring Investigational Site, Montpellier
  - Ferring Investigational Site, Paris
- Italy (4):
  - Ferring Investigational Site, Florence
  - Ferring Investigational Site, Milan
  - Ferring Investigational Site, Napoli
  - Ferring Investigational Site, Roma
- Spain (6):
  - Ferring Investigational Site, Alicante
  - Ferring Investigational Site, Barcelona
  - Ferring Investigational Site, Bilbao
  - Ferring Investigational Site, Madrid
  - Ferring Investigational Site, Málaga
  - Ferring Investigational Site, Valladolid
- United Kingdom (2):
  - Ferring Investigational Site, Coventry
  - Ferring Investigational Site, Liverpool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernabeu A, Zajc P, Garcia Sanchez M, Agrawal R, Papaleo E, Jirecek S, Mogelmose S, Jepsen IE, Lobo R. Ovarian stimulation with follitropin delta for in vitro fertilization: a multicentre, randomized, assessor-blind comparison with follitropin alfa using conventional dosing regimens (ADAPT-1 trial). Hum Reprod. 2025 Sep 1;40(9):1660-1670. doi: 10.1093/humrep/deaf119. PMID 40633120

RESULTS

PARTICIPANT FLOW:
Groups:
- REKOVELLE (Follitropin Delta): REKOVELLE (Follitropin Delta): REKOVELLE administered as single daily subcutaneous injections in the abdomen. The starting dose of REKOVELLE was 15 μg fixed for the first four stimulation days. Dose adjustments could be implemented on the day of starting the gonadotropin-releasing hormone (GnRH) antagonist (stimulation day 5 or day 6) or later, could occur no more frequently than every second day. At each dose adjustment, the daily REKOVELLE dose could be increased or decreased by 5 μg based on the subject's response. The minimum REKOVELLE dose was 5 μg and the maximum REKOVELLE was 20 μg. Subjects could be treated for a maximum of 20 days.
- GONAL-F (Follitropin Alfa): GONAL-F (Follitropin Alfa): GONAL-F administered as single daily subcutaneous injections in the abdomen. The starting dose of GONAL-F was 225 IU fixed for the first four stimulation days. Dose adjustments could be implemented on the day of starting the GnRH antagonist (stimulation day 5 or day 6) or later, could occur no more frequently than every second day. At each dose adjustment, the daily GONAL-F dose could be adjusted by 75 IU based on the subject's response. The minimum GONAL-F dose was 75 IU and the maximum GONAL-F dose was 300 IU. Subjects could be treated for a maximum of 20 days.
Period: Overall Study
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Started | 200 | 100
Completed | 196 | 94
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- REKOVELLE (Follitropin Delta): REKOVELLE (Follitropin Delta): REKOVELLE administered as single daily subcutaneous injections in the abdomen. The starting dose of REKOVELLE is 15 μg fixed for the first four stimulation days. Dose adjustments may be implemented on the day of starting the gonadotropin-releasing hormone (GnRH) antagonist (stimulation day 5 or day 6) or later, can occur no more frequently than every second day. At each dose adjustment, the daily REKOVELLE dose can be increased or decreased by 5 μg based on the subject's response. The minimum REKOVELLE dose is 5 μg and the maximum REKOVELLE is 20 μg. Subjects can be treated for a maximum of 20 days.
- GONAL-F (Follitropin Alfa): GONAL-F (Follitropin Alfa): GONAL-F administered as single daily subcutaneous injections in the abdomen. The starting dose of GONAL-F is 225 IU fixed for the first four stimulation days. Dose adjustments may be implemented on the day of starting the GnRH antagonist (stimulation day 5 or day 6) or later, can occur no more frequently than every second day. At each dose adjustment, the daily GONAL-F dose may be adjusted by 75 IU based on the subject's response. The minimum GONAL-F dose is 75 IU and the maximum GONAL-F dose is 300 IU. Subjects can be treated for a maximum of 20 days.
- Total: Total of all reporting groups
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa) | Total
Number analyzed (Participants) | 200 | 100 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (3.8) | 34.5 (3.4) | 34.5 (3.7)
Age, Customized [Count of Participants; unit: Participants]
  <35 Years | 83 | 43 | 126
  35 - 37 Years | 74 | 39 | 113
  38 - 40 Years | 43 | 18 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 100 | 300
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 20 | 47
  Not Hispanic or Latino | 173 | 80 | 253
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 191 | 98 | 289
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 46 | 22 | 68
  Italy | 35 | 15 | 50
  United Kingdom | 29 | 13 | 42
  France | 5 | 3 | 8
  Spain | 85 | 47 | 132

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Description: The number of oocytes retrieved was recorded at the oocyte retrieval visit.
Time Frame: On day of oocyte retrieval (Up to 22 days after start of stimulation)
Measure: Median (Inter-Quartile Range); unit: Oocytes Retrieved
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 200 | 100
Oocytes Retrieved | 9.0 [6.0 to 13.5] | 9.0 [6.5 to 13.0]

2. Secondary Outcome: Number of Follicles (Total) at End-of-stimulation
Description: Counted by transvaginal ultrasound for the right and left ovary for each subject.
Time Frame: At end-of-stimulation (up to 20 stimulation days)
Measure: Median (Inter-Quartile Range); unit: Follicles
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 200 | 100
Follicles | 12.0 [9.0 to 16.0] | 12.0 [9.0 to 16.0]

3. Secondary Outcome: Size of the Follicles at End-of-stimulation
Description: Counted by ultrasound for the right and left ovary for each subject.
Time Frame: At end-of-stimulation (up to 20 stimulation days)
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 200 | 99
mm | 15.7 [14.7 to 16.8] | 16.0 [15.1 to 16.9]

4. Secondary Outcome: Serum Concentrations of Estradiol at End-of-stimulation
Description: Blood samples for analysis of circulating concentrations of estradiol were drawn.
Time Frame: At end-of-stimulation (up to 20 stimulation days)
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 197 | 96
pmol/L | 6085.0 [3516.0 to 8602.0] | 5853.5 [4053.5 to 9742.0]

5. Secondary Outcome: Serum Concentrations of Progesterone at End-of-stimulation
Description: Blood samples for analysis of circulating concentrations of progesterone were drawn.
Time Frame: At end-of-stimulation (up to 20 stimulation days)
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 197 | 96
nmol/L | 2.9 [1.9 to 3.8] | 2.5 [1.6 to 3.5]

6. Secondary Outcome: Number of Fertilized Oocytes
Description: The number of pronuclei were counted after insemination. Fertilized oocytes with 2 pronuclei (2PN) were regarded as correctly fertilized.
Time Frame: On day 1 after oocyte retrieval (up to 23 days after start of stimulation)
Measure: Median (Inter-Quartile Range); unit: Oocytes
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 200 | 100
Oocytes | 5.0 [3.0 to 8.0] | 5.0 [3.0 to 7.0]

7. Secondary Outcome: Fertilization Rate
Description: The fertilization rate was defined as the number of oocytes with 2PN divided by the number of oocytes retrieved.
Time Frame: On day 1 after oocyte retrieval (up to 23 days after start of stimulation)
Measure: Median (Inter-Quartile Range); unit: percentage of oocytes fertilised
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 198 | 96
percentage of oocytes fertilised | 54.5 [40.0 to 71.4] | 57.7 [40.0 to 71.4]

8. Secondary Outcome: Number of Blastocysts and Number of Good Quality Blastocysts
Description: Number of blastocysts and number of good quality blastocysts on Day 5 or 6 were presented. The quality evaluation of blastocysts consisted of assessment of three parameters, as per the Gardner & Schoolcraft system: blastocyst expansion and hatching status (graded: 1-6), inner cell mass (graded: A-D) and trophectoderm (graded: A-D). A good-quality blastocyst was defined as a blastocyst of grade 3BB or higher.
Time Frame: On Day 5 or Day 6 (as applicable) after oocyte retrieval (up to 27 or 28 days after start of stimulation)
Measure: Median (Inter-Quartile Range); unit: Blastocysts
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 200 | 100
Blastocysts
  Number of Blastocysts | 2.0 [1.0 to 5.0] | 3.0 [1.0 to 4.5]
  Number of good quality blastocysts | 2.0 [1.0 to 4.0] | 2.0 [0.0 to 3.0]

9. Secondary Outcome: Total Gonadotropin Dose
Description: Calculated by start dates, end dates and daily dose of investigational medicinal product (IMP).
Time Frame: Up to 20 stimulation days
Measure: Median (Inter-Quartile Range); unit: ug
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 200 | 100
ug | 135 [120.0 to 160.0] | 148.5 [137.5 to 165.0]

10. Secondary Outcome: Number of Stimulation Days
Description: Calculated by start dates and end dates.
Time Frame: Up to 20 stimulation days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 200 | 100
days | 9.0 [8.0 to 10.0] | 9.0 [8.0 to 10.0]

11. Secondary Outcome: Proportion of Subjects With Early Ovarian Hyperstimulation Syndrome (OHSS) (Overall and by Grade) and/or Preventive Interventions for Early OHSS
Description: Early OHSS is defined as OHSS with onset ≤9 days after triggering of final follicular maturation. Classification of grade was according to Golan's classification system, and all OHSS cases were graded as mild, moderate or severe.
Time Frame: Up to 9 days after triggering of final follicular maturation
Measure: Count of Participants; unit: Participants
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
Number analyzed (Participants) | 200 | 100
Participants
  Early OHSS (any grade) | 5 | 3
  Early OHSS (moderate/severe) | 1 | 1
  Early OHSS (any grade) and / or preventative interventions | 33 | 17
  Early OHSS (moderate/severe) and / or preventative interventions | 30 | 16

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | REKOVELLE (Follitropin Delta) | GONAL-F (Follitropin Alfa)
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/200 | 2/100
Other Adverse Events (participants affected / at risk) | 24/200 | 11/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REKOVELLE (Follitropin Delta) (N=200) | GONAL-F (Follitropin Alfa) (N=100)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REKOVELLE (Follitropin Delta) (N=200) | GONAL-F (Follitropin Alfa) (N=100)
Headache (Nervous system disorders) | 23 (27) | 8 (12)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT05263388/Prot_SAP_000.pdf